CLINICAL TRIAL: NCT01043822
Title: Pain and Emotional Expression in Children With Autism or Mental Retardation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Pr Baghdadli, University Hospital Montpellier
Other Study IDs: UF8481
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Autism; Mental Retardation
Keywords: Autism; mental retardation; pain; emotion; sensory profile; children
MeSH Terms: conditions — Autistic Disorder; Intellectual Disability; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe facial, behavioral and physiologic (heart rate) reactivity of children with autism aged 3 to 6 years old, during a painful stimulation (venepuncture). Children will be videotaped before, during and after a venepuncture. Each recording will be rated with the FACS (Facial Action Coding System) and the NCCPC (Non Communicating Children's Pain Checklist).

DETAILED DESCRIPTION:
Children with autism will be matched with children with mental retardation and children without developmental disorder. Matching will be established according the developmental age of children with autism.

ELIGIBILITY:
Inclusion Criteria:

Group Autism:

* Child aged 3 to 6 years old
* Diagnosis of autistic disorder established according a pluridisciplinary staff (ICD-10 criteria, Vineland scales, ADOS, etc.)
* Admitted to children's neuropediatrics or genetics department for a venepuncture

Control group mental retardation:

* Child aged 3 to 6 years old .
* Diagnosis of mental retardation established according a pluridisciplinary staff (ICD-10 criteria, Vineland scales, ADOS, etc.)
* Admitted to neuropediatric or genetic department for a venepuncture

Control group without developmental disorder :

* Child aged 18 months to 5 years old.
* Admitted to pediatrics department for a venepuncture

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 46 children with autism spectrum disorders, 46 children with mental retardation, 46 children without developmental disorder
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amaria BAGHDADLI, Pr, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France